CLINICAL TRIAL: NCT03273543
Title: Premaxillary Injection for Perioral Rejuvenation and Upper Lip Enhancement
Brief Title: Perioral Rejuvenation and Upper Lip Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Principal Investigator, Steven H. Dayan, MD, FACS, DeNova Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REST-DEF-2017
Record Dates: First submitted 2017-08-30; First posted 2017-09-06 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Perioral Rejuvenation; Upper Lip Projection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Nasal Tip Projection (Experimental)
  Interventions: Device: Restylane® Defyne
- Upper Lip Position (Experimental)
  Interventions: Device: Restylane® Defyne

INTERVENTIONS:
Device: Restylane® Defyne — hyaluronic acid filler injection

SUMMARY:
To determine if subjects who receive premaxillary injection demonstrate an increase in nasal tip projection and an associated increase in upper lip projection, and vermillion height.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects Age 21 to 70. 2. Subjects who demonstrate signs of perioral aging or poor upper lip projection.

Exclusion Criteria:

* 1. Subjects who plan to undergo peri oral neurotoxin treatments or ablative skin treatments, or have had either of these treatments in the previous 6 months, other injectable filler treatments during the course of the study.

  2. Subjects who are pregnant or nursing. 3. Subjects with a known allergy or sensitivity to any component of the study ingredients.

  4. Any history of rhinoplasty or nasal filler injections. 5. Recent history of upper lip augmentation (surgical and non-surgical) within the last 12 months.

  6. Any history of lip lift or other surgical procedures involving the upper lip.

  7. Any history of chin augmentation (surgical and non-surgical). 8. Any history of orthognathic surgery. 9. Any history of bleeding disorders (iatrogenic or otherwise). 10. Current history of chronic drug or alcohol abuse. 11. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study product (i.e. immunosuppressive therapy).

  12. Subjects who, in the Investigator's opinion, have a history of poor cooperation, non¬compliance with medical treatment or unreliability.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Tip Projection | Upper Lip Position
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Tip Projection | Upper Lip Position | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (0) | 41.2 (0) | 39 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Nasal Tip Projection
Description: Baseline nasal projection measurements will be documented according to Goode's ratio.
  The Goode ratio was used as a measurement of tip projection and is defined as the ratio of the nasal height in relation to the nasal length. For each subject's right lateral view photograph, the nasal height was measured as the length of a line drawn from the alar-facial groove to the tip-defining point, and the nasal length was measured as the length of the line drawn from the nasion to the tip-defining point. The nasal height value was then divided by the nasal length value to determine the Goode ratio for a given photograph.
  The ratio of the line from the alar crease to the nasal tip to the nasion to the nasal tip should be . 55. If it is more than that the nose is overprojected, if it is under that ratio the nose is underprojected.
Time Frame: Baseline and 2 months
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Nasal Tip Projection: Restylane® Defyne: hyaluronic acid filler injection
  Mean nasal tip projection measured by comparing baseline vs post-tx Goode's Ratio
Arm/Group | Nasal Tip Projection
Number analyzed (Participants) | 10
ratio | 0.601 (0.052)

2. Primary Outcome: Upper Lip Projection
Description: baseline upper lip position will recorded by measuring the Z-angle, which is the intersection of the Frankfort horizontal line and the profile line as described by Merrifield. From the straight portrait image, the ratio of the upper lip vermillion height to the lower lip vermillion height will be documented.
  Upper lip projection was assessed via measurement of the Z angle. On each subject's right lateral view photograph, a profile line was drawn tangential to the pogonion of the chin and to the most anterior point of the upper lip. A second line was drawn along the Frankfort horizontal plane. The resulting angle at which these two lines intersected corresponded to the Z angle. A decrease in the Z angle to a more acute value on post-treatment photographs would correspond to an increase in upper lip projection.
Time Frame: Baseline and 2 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Upper Lip Position
Number analyzed (Participants) | 10
degrees | 74.245 (10.859)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Nasal Tip Projection | Upper Lip Position
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03273543/Prot_SAP_000.pdf